CLINICAL TRIAL: NCT05810441
Title: Use of Intestinal Transglutaminase Antibodies in the Diagnosis of Celiac Disease in Children and Adults: a Multicenter Prospective Study
Brief Title: Intestinal Transglutaminase Antibodies in Celiac Disease Diagnosis
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 04/19
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Celiac Disease
Keywords: Celiac disease,; Mucosal anti-ttg; Intestinal biopsy culture
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Intestinal biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Typical celiac disease: * symptomatic subjects (gastro-intestinal or extra-intestinal symptoms) tested positive for serum anti-ttg concentrations and with pathological intestinal biopsy;
  * symptomatic and asymptomatic subjects at risk of CD (first-degree relatives of CD patients or subjects with autoimmune disorders) tested positive serum CD antibodies and with atrophic intestinal mucosa
  Interventions: Other: Evaluation of diagnostic accuracy of anti-ttg-m
- Potential celiac disease: Symptomatic subjects tested positive for both serum CD antibodies and anti-ttg-m but with normal intestinal mucosa
  Interventions: Other: Evaluation of diagnostic accuracy of anti-ttg-m
- Control group: Adult and pediatric subjects with inflammatory gastro-intestinal disorders (Crohn disease and ulcerative colitis in acute phase or in remission), oncologic diseases (tumors of the gastro intestinal tract) and infectious diseases (eg Helicobacter pylori gastritis) tested negative for serum anti-ttg
  Interventions: Other: Evaluation of diagnostic accuracy of anti-ttg-m

INTERVENTIONS:
Other: Evaluation of diagnostic accuracy of anti-ttg-m — Mucosal anti-ttg evaluated in intestinal biopsy samples

SUMMARY:
Celiac disease (CD) is a systemic autoimmune gluten-dependent enteropathy in subjects with HLA DQ2/8. CD prevalence is more than 1% with a progression to 2% in adulthood. Among the group at risk such as first-degree relatives, subjects with autoimmune diseases (eg type 1 diabetes) or with syndromes (Down's disease, Turner) the prevalence reaches 5-8%. Recently, in pediatrics CD diagnostic criteria have been modified and the intestinal biopsy can be omitted in presence of a specific clinical and laboratory picture. In the remaining pediatric cases and in all adult patients, the biopsy is fundamental for the diagnosis. The clinical manifestation of CD not always depends on the enteropathy and on the related symptoms, but it can be characterized by extra-intestinal symptoms (eg chronic fatigue, anemia, arthralgia, cerebellar ataxia, alterations of dental enamel) that often hamper a rapid CD recognition delaying the diagnosis especially in adults. Symptoms are not always related to intestinal injury and may be present even when intestinal mucosa is normal. This condition is known as potential CD in which serum IgA anti-transglutaminase antibodies (anti-ttg) are generally positive at low concentrations (eg higher 2-3 times than the cut-off) or positive occasionally. In this clinical context, the gluten-free diet is an effective therapy able to improve the clinical picture and to stop the anti-ttg production. Recent observations, especially in pediatric field, have shown that in potential CD the immunological analysis of intestinal biopsies is characterized by the presence of anti-ttg deposits in the intestinal mucosa which predict the development of intestinal atrophy in a time span of 3- 5 years. Furthermore, these deposits disappear with the diet-therapy. In pediatric field, the diagnostic specificity of mucosal anti-ttg (anti-ttg-m) is between 95-98%, while the sensitivity is 100%. In adults, anti-ttg-m show 100% sensitivity in typical celiac disease (characterized by high serum anti-ttg concentrations and intestinal mucosa atrophy), while no results are available about potential celiac disease. Moreover, in adults data about the specificity of anti-ttg-m in infectious, oncological and inflammatory diseases of the gastro-intestinal tract are not available. The main study objectives are to evaluate anti-ttg-m sensitivity in patients with typical celiac disease and anti-ttg-m specificity in patients with oncological and inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult subjects
* Subjects with clinical suspicion of CD, positive serum anti-ttg concentrations with any value or type of presentation (permanent or fluctuating)
* Asymptomatic or pauci-symptomatic subjects tested positive for serum anti-ttg antibodies during screening test because at risk of CD (eg family members of CD patients, subjects with autoimmune diseases)
* Subjects undergoing gastro-intestinal endoscopy for infectious (eg Helicobacter pylori gastritis), oncologic (tumors of the gastro intestinal tract) or inflammatory disorders (Crohn disease, ulcerative colitis, eosinophilic esophagitis) in acute phase or in remission

Exclusion Criteria:

* Subjects in whom to take biopsies is not indicated during the gastro-intestinal endoscopy
* Subjects with oncological pathology undergoing chemotherapy treatment because anti-blastic agents may play an inhibitory activity in the production of immunoglobulins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult subject. Subjects with clinical suspicion of CD; asymptomatic or pauci-symptomatic subjects tested positive for serum anti-ttg antibodies during screening test because at risk of CD; subjects undergoing gastro-intestinal endoscopy for infectious, oncologic or inflammatory disorders
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the sensitivity of anti-ttg-m for the diagnosis of typical celiac disease in adult and pediatric subjects | At the time of intestinal biopsy
  Anti-ttg-m will be evaluated using direct immunofluorescence and biopsy culture assays. For direct immunofluorescence technique: cryosections of intestinal tissue will be incubated with anti-ttg antibody labeled with rhodamine and subsequently with an antibody against human IgA conjugated with fluorescein. The cryosections will be analyzed with a fluorescence microscope equipped with a software to localize the overlap between red (rhodamine) and green (fluorescein) signals of the two antibodies. For intestinal biopsy culture: biopsies will be maintained in culture medium for 72 hours at 37 °C in the presence of soluble gliadin fragments. After 72 hours the culture liquid will be centrifuged and analyzed for the presence of anti-ttg and anti-endomysium by means of ELISA immuno-enzymatic technique and indirect immunofluorescence assay, respectively. Sensitivity will be evaluated in subjects with typical celiac disease
To evaluate the specificity of anti-ttg-m in the control group | At the time of intestinal biopsy
  Anti-ttg-m will be evaluated as described in Outcome 1. Evaluation of specificity will be carried out in subjects with inflammatory diseases (Crohn disease, ulcerative colitis, in acute phase or in remission) or with oncological pathology at gastro-intestinal level or with infectious disease (Helicobacter pylori) tested negative for serum anti-ttg

SECONDARY OUTCOMES:
To compare immunofluorescence technique and biopsy culture assay in searching anti-ttg-m | At the time of intestinal biopsy
  Anti-ttg-m will be evaluated as described in Outcome 1. Results from immunofluorescence technique and biopsy culture assay will be compared.
To demonstrate the gluten-dependence of anti-ttg-m in potential CD patients by searching anti-ttg-m after gluten-free diet | After 12 months of gluten-free diet
  Anti-ttg-m will be evaluated as described in Outcome 1 in a second biopsy after a period of gluten-free diet

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Zanchi, MD, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS materno infantile Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided